CLINICAL TRIAL: NCT06277440
Title: Cognitive Training Effects for Preschool Children With Attention Deficit Hyperactivity Disorder and Developmental Delays
Brief Title: Cognitive Training for Attention Deficit Hyperactivity Disorder and Developmental Delays
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSTC 112-2314-B-341-001
Record Dates: First submitted 2024-01-05; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Attention Deficit Hyperactivity Disorders; Developmental Delays
Keywords: preschool children; developmental delay; cognitive training; attention deficit hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Twenty preschool children with Attention Deficit Hyperactivity Disorder and developmental delays under rehabilitation therapy will be collected. They will be randomly assigned to the experimental group (receiving rehabilitation therapy and three times per week for 15 minutes, a total of 12 weeks of interactive cognitive training) and the control group (receiving rehabilitation therapy only). Therapeutic effects will be evaluated by an investigator blinded to the group's allocation before and after 12 weeks of treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcome measurements will be performed by a researcher who is blind to the groups' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Traditional rehabilitation program with additional cognitive training
  Interventions: Other: cognitive training
- Active Control (Other): Traditional rehabilitation programs without additional cognitive training
  Interventions: Other: active control

INTERVENTIONS:
Other: cognitive training — cognitive training, 15 min, three times per week, for 12 weeks
  Other Names: traditional rehabilitation programs
  Arms: Intervention group
Other: active control — Traditional rehabilitation programs
  Other Names: traditional rehabilitation programs
  Arms: Active Control

SUMMARY:
To explore whether children with Attention Deficit Hyperactivity Disorder and developmental delays who receive cognitive training and conventional rehabilitation can improve executive function more than traditional rehabilitation alone. A magnetoencephalographic examination will be arranged to explore how brain network activation works.

Research method: 20 preschool children with Attention Deficit Hyperactivity Disorder and developmental delays under rehabilitation therapy will be collected. They will be randomly assigned to the experimental group (receiving rehabilitation therapy and three times per week for 15 minutes, a total of 12 weeks of interactive cognitive training) and the control group (receiving rehabilitation therapy only). Therapeutic effects will be evaluated.

DETAILED DESCRIPTION:
Research method: 20 preschool children with Attention Deficit Hyperactivity Disorder and developmental delays under rehabilitation therapy will be collected. They will be randomly assigned to the experimental group (receiving rehabilitation therapy and three times per week for 15 minutes, a total of 12 weeks of interactive cognitive training) and the control group (receiving rehabilitation therapy only). Therapeutic effects will be evaluated, including Sensory Profile, Swanson, Nolan and Pelham version IV, Conners Kiddie Continuous Performance test, Chinese Childhood Executive Functioning Inventory, and Chinese version of Wechsler Intelligence Scale for Children-IV; and physical health conditions, including Pediatric Daily Occupation Scale, Pediatric Outcome Data Collection Instrument (PODCI), Child Health Questionnaire- Parent Form, Pediatric Quality of Life Inventory (PedsQL)will be evaluated by an investigator who is blinded to the group's allocation at before treatment and after 12 weeks of treatment. All participants will be investigated by magnetoencephalography (MEG) to identify the brain network connectivity while performing different tasks before and after 12 weeks of treatment. Brain Magnetic Resonance Imaging will be performed for brain mapping.

Possible results: The study will shed light on therapeutic effects and brain network connectivity by cognitive training for preschool children with Attention Deficit Hyperactivity Disorder and developmental delays.

ELIGIBILITY:
Inclusion Criteria:

* preschool children with Attention Deficit Hyperactivity Disorder and developmental delays under regular rehabilitation programs intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 4 or greater than 6 metal in teeth intelligence quotient less than 70

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes of executive function | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by the Taiwanese Traditional Chinese Childhood Executive Functioning Inventory range from 1 to 5, higher scores indicate a worse outcome

SECONDARY OUTCOMES:
changes of symptoms of attention deficit hyperactivity disorder | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Swanson, Nolan and Pelham questionnaire, range from 0 to 54, higher scores indicate a worse outcome
changes of attention | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Conners Kiddie Continous Performance Test, range from 0-100, higher scores indicate a worse outcome
Changes of sensory integration | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Sensory Profile, range from 0-100, higher scores indicate a better outcome
changes of intelligence | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by the Wechsler Intelligence Scale of children, the average score is 100, with a higher score indicating higher intelligence and a lower score indicating a lower level of intelligence.
changes of functional performance | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Pediatric Outcome Data Collection Instrument, range from 0-100, higher scores indicate a better outcome
Changes of family impact | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Child Health Questionaire, parent form 28, range from 0-100, higher scores indicate a better outcome
Changes of quality of life | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Pediatric Quality of Life Inventory, range from 0-100, higher scores indicate a better outcome
Changes in performance activity in kindergarten | score change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes in scores assessed by Kindergarten Performance Activity, range from 0-100, higher scores indicate a worse outcome

OTHER OUTCOMES:
changes of brain network connectivity | connectivity change from baseline to 12 weeks of treatment, higher score, the better outcome
  Changes of brain network connectivity assessed by magnetoencephalography, range from 0-1, higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No